CLINICAL TRIAL: NCT00932620
Title: THE EFFECT OF SIMVASTATIN VERSUS COMBINED SIMVASTATIN/EZETIMIBE TREATMENT ON THE CONCENTRATION OF SMALL DENSE LOW-DENSITY LIPOPROTEIN PARTICLES IN PATIENTS WITH PRIMARY HYPERCHOLESTEROLEMIA
Brief Title: Comparison of Simvastatin Versus Simvastatin/Ezetimibe on Small Dense Low -Density Lipoprotein (LDL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Prof. M. Elisaf, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Results first posted 2011-08-12 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-06

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; statins; simvastatin; ezetimibe; LDL particles
MeSH Terms: conditions — Hypercholesterolemia | interventions — Simvastatin; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin 40 mg (Active Comparator): All subjects will receive dietary instructions according to NCEP-ATP III by a clinical nutritionist. If LDL-C is still above recommended levels after 3 months of appropriate lifestyle changes, patients will be randomly allocated to open-label simvastatin 40 mg (n=50) or simvastatin/ezetimibe 10/10 mg (n=50) daily
  Interventions: Drug: SIMVASTATIN 40 mg
- Simvastatin 10 mg plus ezetimibe 10 mg (Active Comparator): All subjects will receive dietary instructions according to NCEP-ATP III by a clinical nutritionist. If LDL-C is still above recommended levels after 3 months of appropriate lifestyle changes, patients will be randomly allocated to open-label simvastatin 40 mg (n=50) or simvastatin/ezetimibe 10/10 mg (n=50) daily
  Interventions: Drug: SIMVASTATIN/EZETIMIBE 10/10 mg

INTERVENTIONS:
Drug: SIMVASTATIN 40 mg — SIMVASTATIN 40 mg/day for 3 months
  Arms: Simvastatin 40 mg
Drug: SIMVASTATIN/EZETIMIBE 10/10 mg — SIMVASTATIN/EZETIMIBE 10/10 mg/day for 3 months
  Arms: Simvastatin 10 mg plus ezetimibe 10 mg

SUMMARY:
Both simvastatin 40 mg and simvastatin/ezetimibe 10/10 mg result in low-density lipoprotein cholesterol (LDL-C) reductions of approximately the same magnitude. However, the differential effects of these two treatment options on small dense LDL-C (sdLDL-C) concentration have not been assessed.

The aim of the present study is to compare the effects of simvastatin 40 mg versus simvastatin/ezetimibe 10/10 mg on sdLDL-C concentration. The primary efficacy endpoint will be changes in LDL subfraction profile (i.e. mean LDL particle size, sdLDL-C levels) at 3 months after treatment initiation.

DETAILED DESCRIPTION:
Hypercholesterolemia is a major risk factor for atherosclerosis and coronary heart disease (CHD).[1] Epidemiological and clinical studies have demonstrated that aggressive lowering of low-density lipoprotein cholesterol (LDL-C) reduces morbidity and mortality in patients with or without CHD.[1-3] LDL consists of an heterogeneous population of particles with respect to size, density and chemical composition. Several studies have shown that small, dense LDL (sdLDL) particles are more atherogenic than large, buoyant ones[4, 5] and thus associated with increased risk for coronary artery disease[6] or stroke.[7] Statins, the mainstay of lipid lowering therapy, achieve significant reductions in LDL-C levels and are suggested to lower all LDL subfractions, possibly as a result of the statin-induced stimulation of LDL-receptor-mediated catabolism.[8] Moreover, several studies have shown that abnormalities in LDL subfraction profile are amenable to correction with statins.[9] Ezetimibe monotherapy has also been found to significantly reduce concentrations of all LDL subfractions.[10] The combination of ezetimibe with low dose of a statin results in similar LDL-C lowering compared with high dose of the same statin. A recent study demonstrated that ezetimibe/simvastatin combination was more effective than ezetimibe and simvastatin monotherapy in reducing atherogenic lipoprotein subfractions in patients with primary hypercholesterolemia.[11] However, in this study ezetimibe/simvastatin combination was more potent in reducing LDL-C levels compared with either monotherapy.[11] In another study, the addition of ezetimibe in patients already receiving atorvastatin decreased LDL-C values exclusively by reducing the concentrations of large, buoyant LDL subfractions.[12] It is so far unknown whether high-dose of a statin would reduce sdLDL-C level more than low-dose statin plus ezetimibe therapy for the same degree of LDL-C lowering.

Both simvastatin 40 mg and simvastatin/ezetimibe 10/10 mg result in LDL-C reductions of approximately the same magnitude.[13,14] However, the differential effects of these two treatment options on sdLDL-C concentration have not been assessed.

Study design Randomized, open label study.

Aim of the study The aim of the present study is to compare the effects of simvastatin 40 mg versus simvastatin/ezetimibe 10/10 mg on sdLDL-C concentration.

Materials and Methods Study population Consecutive patients with primary hypercholesterolemia (n=100) attending the Outpatient Lipid and Obesity Clinic of the University Hospital of Ioannina, Ioannina, Greece will participate in the present study.

All subjects will receive dietary instructions according to National Cholesterol Education Program Adult Treatment Panel III (NCEP-ATP III) by a clinical nutritionist. If LDL-C is still above recommended levels after 3 months of appropriate lifestyle changes, patients will be randomly allocated to open-label simvastatin 40 mg (n=50) or simvastatin/ezetimibe 10/10 mg (n=50) daily.

Enrollment will be completed in a period of 1 year. Follow-up visit will be scheduled at 3 months after treatment initiation.

The study protocol will be approved by the Ethics Committee of the University Hospital of Ioannina and all participants will be asked to give their written informed consent.

Laboratory measurements

Blood analyses will be carried out after an overnight fast (12 hours) and will include:

* Glucose, insulin, creatinine, uric acid, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transpeptidase (γ-GT), alkaline phosphatase (ALP)
* Total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C) and triglyceride levels, whereas LDL-C levels will be assessed using the Friedewald equation (LDL-C = TC-HDL-C-triglycerides/5)
* high-sensitivity C-reaction protein (hs-CRP) levels
* Apolipoproteins A-I, A-II, A-V, B, E, C-II, C-III, lipoprotein (a)[Lp(a)]
* Lipoprotein-associated phospholipase A2 (Lp-PLA2) activity in plasma

Methods LDL subclass analysis Electrophoresis will be performed using high resolution 3% polyacrylamide tube gel and the Lipoprint LDL System (Quantimetrix, Redondo Beach, CA) according to the manufacturer's instructions.[16, 17, 18] Briefly, 25 μl of sample will be mixed with 200 μl of Lipoprint Loading Gel and placed upon the upper part of the 3% polyacrylamide gel. After 30 min of photopolymerization at room temperature, electrophoresis will be performed for 60 min with 3 mA for each gel tube. Each electrophoresis chamber will involve 2 quality controls (sample provided by the manufacturer). For quantification, scanning will be performed with a ScanMaker 8700 digital scanner (Mikrotek Co, USA) and iMac personal computer (Apple Computer Inc, USA). After scanning, electrophoretic mobility (Rf) and the area under the curve (AUC) will be calculated qualitatively and quantitatively with the Lipoprint LDL system Template and the Lipoware software (Quantimetrix Co, Redondo Beach, CA), respectively. The LDL subfraction will be calculated using the Rf between the very low-density lipoprotein (VLDL) fraction (Rf 0.0) and the HDL fraction (Rf 1.0). LDL is distributed from Rf 0.32 to Rf 0.64 as 7 bands, whose Rfs are 0.32, 0.38, 0.45, 0.51, 0.56, 0.6 and 0.64 (LDL1 to LDL7, respectively). LDL1 and LDL2 are defined as large, buoyant LDL and LDL3 to LDL7 are defined as sd-LDL. The cholesterol concentration (in mg/dl) of each LDL subfraction is determined by multiplying the relative AUC of each subfraction by the TC concentration of the sample (the TC concentration of the sample is measured independently). The proportion of sd-LDL-cholesterol (sd-LDL%) will be defined as the percentage of the LDL-cholesterol carried in sd-LDL (i.e. bands 3 to 7). LDL peak particle diameter (LDL-PPD) (nm) will be determined using the Rf of the highest peak of the LDL bands according to the following equation proposed: LDL-PPD = (1.429-Rf)*25. Moreover, the Lipoprint LDL System provides a mean LDL particle size (nm) and uses a size of 26.8 nm as a cut-off point to classify individuals into phenotypes A (absence of sd-LDL particles) and non-A (presence of sd-LDL particles).

Measurement of plasma Lp-PLA2 activity Lp-PLA2 activity in total plasma, in apo B-depleted plasma, after the sedimentation of all apo B-containing lipoproteins with dextran sulfate-magnesium chloride (HDL-Lp-PLA2 activity) as well as in lipoprotein subfractions, will be determined by the trichloroacetic acid precipitation procedure using [3H]-platelet-activating factor (PAF) (100 μM final concentration) as a substrate.[16] The reaction will be performed for 10 min at 37°C and Lp-PLA2 activity will be expressed as nmol PAF degraded per min per ml of plasma or mg of LDL subfraction protein. The non-HDL-Lp-PLA2 activity will be calculated by subtracting the HDL-Lp-PLA2 activity from the total plasma enzyme activity. Lp-PLA2 specific activity will be expressed as a ratio of the enzyme activity to the enzyme mass (nmol/ng/min).

Serum apolipoproteins measurement Serum apolipoproteins A-I, A-II, AV, B, E, C-II, C-III and Lp(a) will be measured by immunonephelometry on a Behring Nephelometer BN ProSpec (Dade-Behring, Lieberbach, Germany).

Determination of plasma hs-CRP levels Plasma concentrations of CRP will be measured with a high sensitivity immunonephelometric assay (Beckman Instruments, Fullerton, CA). The reference range of this assay is 1.0 to 80 mg/l. The detection limit is 1.0 mg/l.

Routine laboratory determinations Routine laboratory determinations will be carried out by automated chemical analysis in the laboratory of the University Hospital of Ioannina using an Olympus AU 600 analyzer (Olympus Diagnostica GmbH, Hamburg, Germany). Glucose will be measured by the hexokinase method and serum insulin levels by the AxSYM Insulin assay, which is based on the Microparticle Enzyme Immunoassay technology (Abbott Laboratories, Diagnostic Division, Abbott Park, IL, USA).

Statistical analysis All parameters will be checked for normality with the Kolmogorov-Smirnov test and non-normal-distributed variables will be log-transformed. Linear regression analysis will be used for the assessment of the relationships between study variables, whereas multivariate analysis will be used for the determination of the independent predictors of study parameter change. The paired-samples t-test will be used for assessing the effect of treatment in each group. Analysis of covariance (ANOVA), adjusted for baseline values, will be used for comparisons between treatment groups. Significance will be defined as p<0.05 and Bonferroni correction will be applied in the case of multiple comparisons. All analyses will be carried out with SPSS 13.0 (SPSS Inc., 1989-2004, Chicago, IL). It was estimated that a sample size of 90 would give a 94% power to detect a 15% difference in the reduction of sdLDL-C concentration between the 2 groups at a 2-sided alpha of 0.05. We will include 100 patients allowing for a drop-out rate of ~10%.

ELIGIBILITY:
Inclusion Criteria:

* LDL-C levels above those recommended by the National Cholesterol Education
* Program Adult Treatment Panel III (NCEP-ATP III) based on each patient risk factors following a 3-month period of lifestyle changes.

Exclusion Criteria:

* Triglycerides >500 mg/dL, renal disease (serum creatinine levels >1.6 mg/dL), hypothyroidism [thyroid stimulating hormone (TSH) >5 IU/mL] and liver disease (ALT and/or AST levels >3-fold upper limit of normal in 2 consecutive measurements).
* Patients with hypertension will be included in the study if they are on stable medication for at least 3 months and their blood pressure is adequately controlled (no change in their treatment will be made during the study period).
* Patients currently taking lipid lowering drugs or having stopped them less than 4 weeks before study entry will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ioannina, Ioannina, Ioannina, Greece

REFERENCES:
- [Result] Florentin M, Liberopoulos EN, Moutzouri E, Rizos CV, Tselepis AD, Elisaf MS. The effect of simvastatin alone versus simvastatin plus ezetimibe on the concentration of small dense low-density lipoprotein cholesterol in subjects with primary hypercholesterolemia. Curr Med Res Opin. 2011 Mar;27(3):685-92. doi: 10.1185/03007995.2010.546394. Epub 2011 Jan 27. PMID 21271793
- See also: 2nd Department of Internal Medicine, University Hospital of Ioannina — http://www.bpath.gr

RESULTS

PARTICIPANT FLOW:
Groups:
- Simvastatin 40 mg: All subjects will receive dietary instructions according to NCEP-ATP III by a clinical nutritionist. If LDL-C is still above recommended levels after 3 months of appropriate lifestyle changes, patients will be randomly allocated to open-label simvastatin 40 mg daily
- Simvastatin 10 mg Plus Ezetimibe 10 mg: All subjects will receive dietary instructions according to NCEP-ATP III by a clinical nutritionist. If LDL-C is still above recommended levels after 3 months of appropriate lifestyle changes, patients will be randomly allocated to open-label simvastatin/ezetimibe 10/10 mg (n=50) daily
Period: Overall Study
Arm/Group | Simvastatin 40 mg | Simvastatin 10 mg Plus Ezetimibe 10 mg
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin 40 mg | Simvastatin 10 mg Plus Ezetimibe 10 mg | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 44 | 89
  >=65 years | 5 | 6 | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 57 (10) | 59 (9) | 58 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 34 | 33 | 67
Region of Enrollment [Number; unit: participants]
  Greece | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Changes in Small Dense Low-density Lipoprotein Cholesterol (sdLDL-C) Levels
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: sdLDL-C, mg/dL
Arm/Group | Simvastatin 40 mg | Simvastatin 10 mg Plus Ezetimibe 10 mg
Number analyzed (Participants) | 50 | 50
sdLDL-C, mg/dL | -42 (10) | -46 (13)

2. Secondary Outcome: Changes in Low-density Lipoprotein Cholesterol (LDL-C)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: LDL-C, mg/dL
Arm/Group | Simvastatin 40 | Simvastatin/Ezetimibe 10/10
Number analyzed (Participants) | 50 | 50
LDL-C, mg/dL | -43 (10) | -49 (12)

ADVERSE EVENTS:
Arm/Group | Simvastatin 40 mg | Simvastatin 10 mg Plus Ezetimibe 10 mg
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
Limitations of our study include its open-label design and the lack of clinical endpoints. However, all laboratory determinations were performed blindly with regard to treatment allocation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No